CLINICAL TRIAL: NCT01685853
Title: Bowel Cleansing for Colonoscopy: Comparison Between a Same Day Low-Volume Preparation and a Conventional 4L Split One. A Randomized, Observer-blind, Parallel Group, Comparative Study.
Brief Title: Bowel Cleansing for Colonoscopy: Comparison Between a Same Day Low-Volume Preparation and a Conventional 4L Split One
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEO S570 510; 2010-022967-37 (EudraCT Number)
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG 4 litres split (Active Comparator): Polyethylene glycol with electrolytes (PEG)
  Interventions: Drug: PEG 4 litres split
- Bisacodyl plus PEG-CS (Experimental): Bisacodyl plus PEG-CS: Bisacodyl plus Polyethylene glycol with citrate and simethicone (PEG-CS)
  Interventions: Drug: Bisacodyl plus PEG-CS

INTERVENTIONS:
Drug: Bisacodyl plus PEG-CS — * the day before colonoscopy: 3-4 bisacodyl tablets (according to patient bowel habit) at bedtime
  * the morning of colonoscopy: PEG-CS (2 litres) starting 5 hours before the exam
  Other Names: LOVOLdyl plus LOVOLesse
  Arms: Bisacodyl plus PEG-CS
Drug: PEG 4 litres split — * the day before colonoscopy: 2 litres of PEG
  * the morning of colonoscopy: 2 litres of PEG starting 5 hours before the examination
  Other Names: SELG 1000
  Arms: PEG 4 litres split

SUMMARY:
The present study is intended to evaluate the effectiveness, tolerability, compliance, and feasibility of the low volume bowel preparation, bisacodyl tablets followed by 2L Polyethylene glycol (PEG) with citrate and simethicone (CS) given the same day of colonoscopy, vs the standard 4L split PEG solution.

DETAILED DESCRIPTION:
Eligible patients will be informed about the aims, procedures, benefits and possible risks of the study prior to sign the informed consent form from day -30 to day-3. They will provide medical history and undergo a physical examination. Patients will be evaluated by a Physician other than the blind Endoscopist. The same responsible person will instruct the patients about administration procedures in both oral and written form. The patients will be assigned to receive one of the dosing schedule bowel preparation according to a computer generated block-randomisation list. Patients will take the study treatment at home according to the given instructions. Patients will return to the clinic for colonoscopy. The colonoscopy will be performed by an Endoscopist who will be unaware of the bowel dose-regimen preparation taken by the patient. Completed colonoscopic exam will be performed with time recorded (intubation and withdrawal from ceacum). The unblind Investigator will ask the patients about safety, tolerability, overall acceptance and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients undergoing a complete colonoscopy
* Patient written informed consent

Exclusion Criteria:

* Pregnant or lactating women or at a risk of becoming pregnant
* Known or suspected gastrointestinal obstruction or perforation; toxic megacolon; major colonic resection Known or suspected hypersensitivity to the active principle and/or formulations' ingredients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | 20 min
  Evaluation of the quality of bowel preparation according to the Ottawa Scale

SECONDARY OUTCOMES:
Efficacy | 20 min
  Evaluation of the mucosal visibility according to a 3 point scale (0-2)
Efficacy | 20 min
  Adenoma detection rate
Safety | 24 hours
  Recording of all adverse events occurred during the study by patient questioning
Tolerability | 24 hours
  rate of patients in the two groups who developed GI symptoms related to bowel preparation
Acceptability | 24 hours
  willingness to repeat the preparation
Compliance | 24 hours
  rate of patient with intake of at least 75% of bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Crosta, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy